CLINICAL TRIAL: NCT04546087
Title: Impact of Labor and Delivery on Ultrasound Measured Cricothyroid Membrane Depth and Height
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-01
Record Dates: First submitted 2020-08-28; First posted 2020-09-11 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Airway Complication of Anesthesia
Keywords: cricothyroid membrane; pregnancy; ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound (Experimental): Ultrasound measurements of the cricothyroid membrane.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound scan of the cricothyroid membrane

SUMMARY:
The cricothyroid membrane acts as a route through which the upper airway can be accessed to provide oxygen and ventilation to patients. Anesthesiologists need to deliver oxygen and ventilation to patients under general anesthesia, where patients may lose the ability to breath for themselves. Access through this membrane to provide oxygen and ventilation is critical in emergency situations where other traditional means to access the airway (e.g. through endotracheal ventilation, supraglottic airway devices or face mask ventilation) have failed. It is known, from previous studies, that due to the physiological changes that occur in labour, the upper airway of the body undergoes changes that can make accessing the airway through traditional means more difficult, specifically during the period of labor, delivery, and just after delivery. Ultrasound is becoming increasingly popular due to its ability both to identify the cricothyroid membrane and to improve success in accessing the airway through the cricothyroid membrane. What is not known, and has not been studied to date, is specifically how the anatomy (i.e. its height and its depth) specifically changes during the period of labour, delivery and just after delivery.

The aim of this study would be to scan (using ultrasound) pregnant women's necks once at the very start of their labour, and once within 4 hours of delivery of their baby, to identify how the size and depth of the cricothyroid membrane changes. This information would improve the understanding of how to best approach accessing this membrane in laboring pregnant women.

The investigators hypothesize that in labouring third trimester patient, that the depth to the cricothyroid membrane will increase, and there will be no change in the cricothyroid membrane height.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years old
* Pregnant patients in third trimester (>28/40 weeks)
* Ability to understand the rationale of the study assessments and to provide signed consent.

Exclusion Criteria:

* Neck arthritis
* Cervical stenosis
* Known cervical degenerative disc disease
* Rheumatoid Arthritis
* Any restriction of neck movement
* Upper limb neurology
* Patient refusal
* Patients not in established labour.
* Patients undergoing cesarean section
* Known distorted airway anatomy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Cricothyroid membrane position change | 24 hours
  Difference between the depth from the skin to the cricothyroid membrane- tracheal interface change ultrasound between the onset of established labor and following delivery of the baby and placenta.

SECONDARY OUTCOMES:
Cricothyroid membrane size change | 24 hours
  Difference between the height of the cricothyroid membrane (CTM) at the onset of established labor and the height of CTM following delivery of the baby.

CONTACTS AND LOCATIONS:
Overall Officials: Eric You-Ten, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No